CLINICAL TRIAL: NCT06335030
Title: Relationship Between Sensory and Behavioral Aspects With Particular Attention to Food Selectivity in Children With Autism Spectrum Disorder and Parental Stress Perceived
Brief Title: Sensory and Behavioral Aspects With Particular Attention to Food Selectivity in Children With Autism
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Ospedale Borgo Trento - Verona (Other); Università degli Studi di Trento (Other)
Responsible Party: Principal Investigator, Raffaella Tancredi, MD Director Clinical Unit, IRCCS Fondazione Stella Maris
Other Study IDs: 2.1_AUT-SP2_001_Tancredi
Record Dates: First submitted 2024-03-04; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Food Selectivity; Autism; Parental Stress; Sensory Profile
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary: Eating problems and in particular food selectivity is a condition that worsens a long-life disorder such as Autism Spectrum Disorder (ASD) , both on an individual level, both on family and social ones .

Children (2-6 years) diagnosed with ASD according to Diagnostic and Statistical Manual of Mental Disorders 5 Edition (DSM5) criteria were enrolled in an observational, cross-sectional and multicentric study conducted by three different Italian clinical centers. Regarding this sample, principal aims of the study are to describe characteristics of food selectivity, to evaluate its correlation with ASD symptoms, with cognitive and adaptive functioning of ASD preschoolers, to describe its impact on parental stress.

DETAILED DESCRIPTION:
Background: Eating problems and in particular food selectivity is a condition that worsens a long-life disorder such as ASD, both on an individual level , both on family and social ones . Regarding factors that contribute to this eating behavior have been identified sensory atypia , rigid behaviors and behavioral problems , however the problem has not yet been fully clarified.

Objective: The study aims to:

a) evaluate the presence and characteristics of food selectivity, in a sample of preschool children with ASD, the impact of this on the child's height and weight growth, the possible correlation with gastrointestinal symptoms and with oro-motor skills; b) assess the correlation between food selectivity and the characteristics of ASD (sensory atypia, repetitive behaviors, level of severity of symptoms), the cognitive development/ability quotient, adaptive functioning and the presence of behavioral disorders; c) highlight the impact of food selectivity of ASD children on parental stress.These aims are relevant in order to identify possible future therapeutic interventions that rate both the child's needs and parents involvement.

Methods: children (2-6 years) diagnosed with ASD according to DSM-5 criteria at the IRCCS Stella Maris institute (Clinical Unit ASD Department), were enrolled in an observational, cross-sectional and multicentric study conducted by three different Italian clinical centers (IRCCS Stella Maris Foundation Pisa, Regional Center for Autism Spectrum Disorders - Verona, Observation Diagnostic Training Lab - Trento). This study received the approval of the Tuscany Regional Ethics Committee for the pediatric age (Meyer).

In detail, the study involves parents by administering an anamnestic interview regarding the medical history and development of the child, the rehabilitation and pharmacological intervention in progress; the collection of a video recording of two meals in a family context. Parents complete a series of questionnaires including Child Oral and Motor Proficiency Scale( ChOMPS ), Brief Autism Mealtime Behavior Inventory, (BAMBI) ; Sensory Profile 2( SP2); Child Behavior Checklist (CBCL) 1.5-5 or 6-18 ; Parenting Stress Index, (PSI); Food diary ; Autism-Spectrum Quotient Test (AQ) ); Gastrointestinal Symptom Severity Index (GISSI); Mac Arthur questionnaire . The study includes the evaluation of children' cognitive functioning through the administration of a psychometric/developmental test, the administration of a standardized test for the evaluation of socio-communicative skills (Autism Diagnostic Observation Schedule 2 Edition ) and the observation of a meal of the child at the institute. The study provides a database dedicated to the collection data obtained.

As regards the statistical analyses, the researchers want to examine subjects affected by food selectivity identified and compared with the remaining group. A clinical characterization of children with food selectivity will be defined to describe any differences in the sensory profile and in eating difficulties based on the characteristics of the ASD and the cognitive abilities of the children. Then the impact of the same eating difficulties will be evaluated on the child's adaptive and emotional difficulties and on parental stress index.

ELIGIBILITY:
Inclusion Criteria

* Children (2-6 years)
* diagnosed with ASD according to DSM-5 criteria at the IRCCS Stella Maris institute (Operational Unit 3 ASD Department)

Exclusion Criteria:

* Brain Malformation
* Genetic syndromes
* specifical neurological signs
* prematurity
* epilepsy
* non free diet.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: children (2-6 years) diagnosed with ASD according to DSM-5 criteria at the IRCCS Stella Maris institute (Operational Unit 3 ASD Department), were enrolled in an observational, cross-sectional and multicentric study conducted by three different Italian clinical centers (IRCCS Fondazione Stella Maris - Pisa, Regional Center for Autism Spectrum Disorders - Verona, ODFLab - Trento).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Child Oral and Motor Proficiency Scale (ChOMPS) | baseline
  It is a questionnaire that evaluates the motor and oral-motor skills that underlie the eating and drinking ability for children aged six months to seven years. It consists of a score total divided into four different subscales: "basic movement patterns", "oral-motor skills fundamentals", "oral-motor coordination" and "complex movement patterns".
Brief Autism Mealtime Behavior Inventory (BAMBI) | baseline
  It is a questionnaire consisting of 15 items for the evaluation of food problems referable to a food selectivity framework (total score greater than or equal to 34). It includes four different domains "food selectivity", "destructive behaviors during meals", "food refusal","rigidity during meals" and a total score.
Sensory Profile 2 (SP2) | baseline
  This questionnaire administered to parents, has the purpose of identifying atypical sensory processing and in particular impairments referable to sensory processing that could be related to food selectivity (normal profile,moderately atypical or clearly atypical for age in the processing of individuals sensory channels, in modulation, in behavior and emotional responses).
Child Behavior Checklist (CBCL) | baseline
  It is used to evaluate developmental psychopathology through scales that assess specific dimensions (Anxiety/Depression; Withdrawal/Depression; Somatic Complaints; Social Problems; Thinking Problems; Attention Problems; Rule-Breaking Behaviors; Aggressive Behaviors), general (Internalizing, Externalizing, and Total Problems), emotional-behavioral problems according to some of the DSM diagnostic categories (Affective Problems; Anxiety Problems; Somatic Problems; Attention-Deficit/Hyperactivity Problems; Oppositional-Provocative Problems; Conduct Problems). In the present study parent form is used.
Parenting Stress Index (PSI) | baseline
  It is a questionnaire that measures parental stress level in the parent-child system. It is made up of two domains, Child Domain and Parent Domain composed by 4 sub-scales, which together form the Total Stress scale.The Short Form of PSI-4 (PSI-4-SF) is organized into three sub-scales, Parental Distress, Parent-Child Interaction dysfunctional and Difficult Child. There is also the Defensive Response, which allows you to have information on the respondent's defensive attitude.
Observation of child meal-time | baseline
  On-line observation of child habits during meal-time
Food Diary | baseline
  It was adapted from the original one of the "Zoom8"survey financed by the Istituto Superiore di Sanità, which studies adherence to the Mediterranean diet in school-age children in Italy. The parents of each child included in the study will record the usual eating habits of his/her child refer to the last year. Its administration has the aim of analyzing the types of foods taken by children with ASD with or without food selectivity
Gastrointestinal severity symptom index (GSSI) | baseline
  It is a questionnaire to evaluate presence of gastrointestinal symptoms. It takes 5-10 minutes to compile. A score of 4 or higher (with at least 3 points deriving from the first 6 items which specifically investigate the most common symptoms gastrointestinal) is considered clinically significant to identify relevant gastrointestinal symptoms. There is also an additional section on behaviors associated (verbal and motor) which have been linked to the presence of gastrointestinal symptoms in subjects with ASD.
Mac Arthur | baseline
  It is a questionnaire to evaluate the linguistic level. It collects important information on the development of children's abilities in language, including receptive vocabulary, production, gestures repertoire and grammar.

SECONDARY OUTCOMES:
Autism Quotient (AQ) | baseline
  It is a questionnaire administered to parents separately to evaluate autism traits.
Autism Diagnostic Observation Schedule-2 (ADOS-2) | baseline
  It is a standardized test for the evaluation of socio-communicative skills. In the present study participants completed the Toddler Module (designed specifically for children 12-30 months old with limited language), the Module 1 (used for children aged from 31 months who do not consistently use phrase speech) or the Module 2 (used for children using phrase speech, but who were not verbally fluent) and Module 3(used for children were verbally fluent). To allow comparisons among different modules, ADOS-2 scores (total score, Social Affect, SA, and Restricted and Repetitive Behaviour, RRB, scores) were converted to respective calibrated severity scores (CSS 1-10 indicating absence to severe autism).
Vineland-II scales (VABS II) | baseline
  It assess adaptive behavior in terms of abilities for personal and social functioning in different domains of everyday life. Each domain comprises subdomains (Receptive, Expressive, and Written skills in Communication; Personal, Domestic, and Community skills of Daily Living; Interpersonal relationship, Play and leisure time, and Coping skills of Socialization; and Gross and Fine Motor skills) with item sets assessing specific content areas. In the present study, the scores obtained Communication, Daily living skills, and Socialization domains were used.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Tancredi, Principal Investigator — IRCCS Stella Maris
Locations (3):
- Italy (3):
  - IRCCS Stella Maris, Pisa, PI
  - Università degli Studi di Trento-Laboratorio di Osservazione, Diagnosi e Formazione, Rovereto
  - Azienda Ospedaliera Borgo Trento, Verona

IPD SHARING:
Plan to Share IPD: Undecided
Local database

REFERENCES:
- [Background] Curtin C, Hubbard K, Anderson SE, Mick E, Must A, Bandini LG. Food selectivity, mealtime behavior problems, spousal stress, and family food choices in children with and without autism spectrum disorder. J Autism Dev Disord. 2015 Oct;45(10):3308-15. doi: 10.1007/s10803-015-2490-x. PMID 26070276
- [Background] Evans EW, Must A, Anderson SE, Curtin C, Scampini R, Maslin M, Bandini L. Dietary Patterns and Body Mass Index in Children with Autism and Typically Developing Children. Res Autism Spectr Disord. 2012;6(1):399-405. doi: 10.1016/j.rasd.2011.06.014. PMID 22936951
- [Background] Johnson CR, Turner K, Stewart PA, Schmidt B, Shui A, Macklin E, Reynolds A, James J, Johnson SL, Manning Courtney P, Hyman SL. Relationships between feeding problems, behavioral characteristics and nutritional quality in children with ASD. J Autism Dev Disord. 2014 Sep;44(9):2175-84. doi: 10.1007/s10803-014-2095-9. PMID 24664635
- [Background] Lukens CT, Linscheid TR. Development and validation of an inventory to assess mealtime behavior problems in children with autism. J Autism Dev Disord. 2008 Feb;38(2):342-52. doi: 10.1007/s10803-007-0401-5. Epub 2007 Jun 20. PMID 17578658
- [Background] Muratori F, Tonacci A, Billeci L, Catalucci T, Igliozzi R, Calderoni S, Narzisi A. Olfactory Processing in Male Children with Autism: Atypical Odor Threshold and Identification. J Autism Dev Disord. 2017 Oct;47(10):3243-3251. doi: 10.1007/s10803-017-3250-x. PMID 28744761
- [Background] Prosperi M, Santocchi E, Balboni G, Narzisi A, Bozza M, Fulceri F, Apicella F, Igliozzi R, Cosenza A, Tancredi R, Calderoni S, Muratori F. Behavioral Phenotype of ASD Preschoolers with Gastrointestinal Symptoms or Food Selectivity. J Autism Dev Disord. 2017 Nov;47(11):3574-3588. doi: 10.1007/s10803-017-3271-5. PMID 28861653
- See also: Description of PSI — https://effectiveservices.my.site.com/s/measure/a007R00000v8QbCQAU/parenting-stress-index
- See also: Description and scoring CBCL — https://aseba.emedea.it/